CLINICAL TRIAL: NCT00747435
Title: The MED-EL EAS (Electric-Acoustic System) Using the PULSARCI100 FLEXeas / SONATATI100 FLEXeas and the DUET Speech Processor
Brief Title: Safety and Effectiveness of the MED-EL Electric-Acoustic System
Acronym: EAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G040002
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Hearing Loss
Keywords: sensorineural hearing loss; ski slope audiogram; electric acoustic stimulation
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Original Audiological Criteria (Experimental): Inclusion Criteria:
  Pure-tone air-conduction threshold levels shall fall at or within the levels listed in the following chart.
  Frequency (Hz): 250 500 750 1000 1500 2000 4000 8000 Lower Limit: 10 10 10 60 60 70 70 70 Upper Limit: 65 65 75 *110+ *110+*110+ *110+ *90+
  Minimal benefit from optimally fit hearing aid/s, preferably bilateral, with monosyllabic word scores in quiet of ≤50% in the best-aided condition.
  Interventions: Device: Electric Acoustic System
- Expanded Audiological Criteria (Experimental): Pure-tone air-conduction threshold levels shall fall at or within the levels listed in the following chart.
  Frequency (Hz): 250 500 750 1000 1500 2000 4000 8000 Lower Limit: 10 10 10 60 60 70 70 70 Upper Limit: 65 65 75 *110+ *110+*110+ *110+ *90+
  Minimal benefit from optimally fit hearing aid/s, preferably bilateral, with monosyllabic word scores in quiet of ≤50% in the best-aided condition.
  Study Arm 2 candidates are those who meet the inclusion criteria listed above with the exception that:
  In the ear to be implanted, the pure-tone air conduction threshold(s) at 250, 500, and/or 750 Hz will be greater than or equal to 0 dB HL and less than 10 dB HL, and/or In the ear to be implanted, the pure-tone air conduction threshold(s) at 1000 and/or 1500 Hz will be greater than or equal to 0 dB HL and less than 60 dB HL and/or In their best-aided condition, they score 51-60% on monosyllabic word scores.
  Interventions: Device: Electric Acoustic System

INTERVENTIONS:
Device: Electric Acoustic System — Combination of a cochlear implant and a hearing aid
  Other Names: EAS; Electric Acoustic Systems

SUMMARY:
The purpose of this investigation is to demonstrate the safety and effectiveness of the MED-EL Electric-Acoustic System (EAS), a medical device that combines the use of a cochlear implant with an external electric-acoustic processor designed to provide benefit in speech perception and sound quality to individuals with a sensorineural hearing loss with minimal changes in residual hearing. The acoustic component of the processor will aid residual acoustic hearing in low frequency ranges, while the cochlear implant and electric component of the processor will be used to electrically stimulate the auditory nerve across a wide range of frequencies necessary for speech perception.

ELIGIBILITY:
Inclusion Criteria:

* Audiologic tests suggest a moderate sloping to severe/profound sensorineural hearing loss in the ear to be implanted. The non-implanted ear may fall outside of these criteria; however, threshold levels cannot be better than the indication criteria (for example, the non-implanted ear must be 60 dB or poorer at 1000 Hz, 70 dB or poorer at 2000-8000 Hz).
* Pure-tone air-conduction threshold levels for the ear to be implanted shall fall at or within the following levels:

  250 Hz - 500 Hz hearing loss less than or equal to 65 dB HL 750 Hz hearing loss less than or equal to 75 dB HL 1000-1500 Hz hearing loss less than or equal to 60 dBHL (ie. 60-110+ dB HL) 2000 Hz - 8000 Hz hearing loss less than or equal to 70 dB HL
* Pure-tone air-conduction threshold levels shall fall at or within the levels listed in the following chart Frequency (Hz): 250 500 750 1000 1500 2000 4000 8000 Lower Limit: 10 10 10 60 60 70 70 70 Upper Limit: 65 65 75 *110+ *110+ *110+ *110+ *90+
* Pure-tone air-conduction thresholds for both ears are within 20 dB of each other at 250, 500 and 1000 Hz.
* Air-bone gap at 500, 1000, 2000 and 4000 Hz should be <10 dB at two or more of these frequencies.
* Minimal benefit from optimally fit hearing aid/s, preferably bilateral, with monosyllabic word scores in quiet of ≤50% in the best-aided condition.
* Normal middle ear anatomy and function (based on clinical assessment of tympanometry and acoustic reflex results). No prior middle ear surgery or history of postadolescent, chronic middle ear infections or inner ear disorders (i.e. vertigo or Meniere's syndrome).
* No evidence that hearing loss origin is retrocochlear.
* Current user of bilateral acoustic hearing aids for at least 3 months. Note: If the subject has not been a successful hearing aid user (i.e. improper fit, feedback and/or discomfort from high frequency amplification), he/she must complete a hearing aid trial in the ear to be implanted for at least 1 month. If the ear to be implanted is poorer than the contralateral ear, then the subject must complete a hearing aid trial in both ears for at least 1 month to ensure that he/she is tested in the best-aided condition.
* Adults 18-70 years of age at time of implantation.
* Persons who currently exhibit sufficient understanding and communicative skills to comprehend general conversation in an "oral/aural mode" through normal conversation channels.
* English as primary language.
* Appropriate motivation and expectation levels.

Expanded Criteria:

Study Arm 2 candidates are those who meet the inclusion criteria listed above with the exception that:

In the ear to be implanted, the pure-tone air conduction threshold(s) at 250, 500, and/or 750 Hz will be greater than or equal to 0 dB HL and less than 10 dB HL, and/or In the ear to be implanted, the pure-tone air conduction threshold(s) at 1000 and/or 1500 Hz will be greater than or equal to 0 dB HL and less than 60 dB HL and/or In their best-aided condition, they score 51-60% on monosyllabic word scores.

Exclusion Criteria:

* Conductive, retrocochlear or central auditory disorders.
* Hearing loss in the ear to be implanted that has demonstrated a recent fluctuation at two or more frequencies of 15 dB in either direction in the last 2 years as demonstrated by serial audiograms. Note: In cases where 2-year documentation is missing, documentation of at least 18 months is necessary along with patient report of no fluctuation in the past 2 years. If 18-month data is unavailable, the patient must be monitored until 18-month data is available.
* Any physical, psychological, or emotional disorder that would interfere with surgery or the ability to perform on test and rehabilitation procedures.
* Developmental delays or organic brain dysfunction.
* Physical or geographic limitations that may interfere with the completion of scheduled follow-up evaluations.
* Skin or scalp conditions that could preclude magnetic attachment of the speech processor or use of the acoustic hearing aid.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Tucci, MD, Principal Investigator — Duke University; Christina Runge, PhD, Principal Investigator — Medical College of Wisconsin; Michael Ruckenstein, MD, Principal Investigator — University of Pennsylvania; Hinrich Staecker, MD, Principal Investigator — University of Kansas Medical Center; Peter Roland, MD, Principal Investigator — University of Texas Southwestern Medical Center; Oliver Adunka, MD, Principal Investigator — University of North Carolina Hospital; Ronald Hoffman, MD, Principal Investigator — New York Eye and Ear; Richard Miyamoto, MD, Principal Investigator — Indiana University School of Medicine; Teresa Zwolan, PhD, Principal Investigator — University of Michigan; Nikolas Blevins, MD, Principal Investigator — Stanford University; Rodney Lusk, MD, Principal Investigator — Boys Town; Fred Telischi, MD, Principal Investigator — University of Miami; Douglas Backous, MD, Principal Investigator — Swedish Medical Center; Frank Warren, MD, Principal Investigator — Oregon Health Sciences Center
Locations (14):
- United States (14):
  - Stanford University Medical Center, Stanford, California
  - University of Miami, Miami, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Boys Town, Omaha, Nebraska
  - New York Eye & Ear, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health Sciences Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Skarzynski H, Lorens A, Piotrowska A, Anderson I. Preservation of low frequency hearing in partial deafness cochlear implantation (PDCI) using the round window surgical approach. Acta Otolaryngol. 2007 Jan;127(1):41-8. doi: 10.1080/00016480500488917. PMID 17364328
- [Background] Skarzynski H, Lorens A, Piotrowska A, Anderson I. Partial deafness cochlear implantation provides benefit to a new population of individuals with hearing loss. Acta Otolaryngol. 2006 Sep;126(9):934-40. doi: 10.1080/00016480600606632. PMID 16864490
- [Background] Skarzynski H, Lorens A, Piotrowska A. [New method of partial deafness treatment]. Otolaryngol Pol. 2004;58(4):811-6. Polish. PMID 15603395
- [Background] Skarzynski H, Lorens A, Piotrowska A. A new method of partial deafness treatment. Med Sci Monit. 2003 Apr;9(4):CS20-4. PMID 12709676
- [Background] Kiefer J, Pok M, Adunka O, Sturzebecher E, Baumgartner W, Schmidt M, Tillein J, Ye Q, Gstoettner W. Combined electric and acoustic stimulation of the auditory system: results of a clinical study. Audiol Neurootol. 2005 May-Jun;10(3):134-44. doi: 10.1159/000084023. Epub 2005 Feb 17. PMID 15724084
- [Background] Kiefer J, Gstoettner W, Baumgartner W, Pok SM, Tillein J, Ye Q, von Ilberg C. Conservation of low-frequency hearing in cochlear implantation. Acta Otolaryngol. 2004 Apr;124(3):272-80. doi: 10.1080/00016480310000755a. PMID 15141755
- [Background] von Ilberg C, Kiefer J, Tillein J, Pfenningdorff T, Hartmann R, Sturzebecher E, Klinke R. Electric-acoustic stimulation of the auditory system. New technology for severe hearing loss. ORL J Otorhinolaryngol Relat Spec. 1999 Nov-Dec;61(6):334-40. doi: 10.1159/000027695. PMID 10545807
- [Background] Gstoettner WK, Helbig S, Maier N, Kiefer J, Radeloff A, Adunka OF. Ipsilateral electric acoustic stimulation of the auditory system: results of long-term hearing preservation. Audiol Neurootol. 2006;11 Suppl 1:49-56. doi: 10.1159/000095614. Epub 2006 Oct 6. PMID 17063011
- [Background] Gstoettner W, Kiefer J, Baumgartner WD, Pok S, Peters S, Adunka O. Hearing preservation in cochlear implantation for electric acoustic stimulation. Acta Otolaryngol. 2004 May;124(4):348-52. doi: 10.1080/00016480410016432. PMID 15224851
- [Result] Gstoettner WK, van de Heyning P, O'Connor AF, Morera C, Sainz M, Vermeire K, Mcdonald S, Cavalle L, Helbig S, Valdecasas JG, Anderson I, Adunka OF. Electric acoustic stimulation of the auditory system: results of a multi-centre investigation. Acta Otolaryngol. 2008 Sep;128(9):968-75. doi: 10.1080/00016480701805471. PMID 19086194

RESULTS

PARTICIPANT FLOW:
Groups:
- Original Audiological Criteria: Originally the study was designed to have two ARMs, but the second study ARM did not fully enroll. At the time of submission, the data for both ARMs was collapsed and data analysis was completed on all subjects as one group. The below inclusion criteria represents both ARMs as one group.
  Inclusion Criteria:
  Pure-tone air-conduction threshold levels shall fall at or within the levels listed in the following chart.
  Frequency (Hz): 250 500 750 1000 1500 2000 4000 8000 Lower Limit: 0 0 0 0 0 70 70 70 Upper Limit: 65 65 75 *110+*110+ *110+ *110+ *90+
  Minimal benefit from optimally fit hearing aid/s, preferably bilateral, with monosyllabic word scores in quiet of ≤60% in the best-aided condition.
  Electric Acoustic System: Combination of a cochlear implant and a hearing aid
Period: Overall Study
Arm/Group | Original Audiological Criteria
Started | 73
Completed | 67
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Still undergoing follow up | 1

BASELINE CHARACTERISTICS:
Population: 6 participants withdrew before study completion, outcome measures are reported 67 participants
Groups:
- Original Audiological Criteria: Inclusion Criteria:
  Pure-tone air-conduction threshold levels shall fall at or within the levels listed in the following chart.
  Frequency (Hz): 250 500 750 1000 1500 2000 4000 8000 Lower Limit: 0 0 0 0 0 70 70 70 Upper Limit: 65 65 75 *110+*110+ *110+ *110+ *90+
  Minimal benefit from optimally fit hearing aid/s, preferably bilateral, with monosyllabic word scores in quiet of ≤60% in the best-aided condition.
  Electric Acoustic System: Combination of a cochlear implant and a hearing aid
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 73
Age, Continuous [Mean (Full Range); unit: years] | 53.7 [17 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 73
Duration of hearing loss [Mean (Full Range); unit: years] | 25.7 [2 to 60]

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Speech Perception in Noise With EAS When Compared to the Preoperative Hearing Aid Alone Condition.
Description: CUNY sentences in noise are scored as the percent correct of words in each sentence. The total percent correct for preoperative hearing aid use was subtracted from the total percent correct for EAS at 12 months giving a percentage point improvement in speech perception with EAS.
Time Frame: 12 months post initial activation
Population: One subject lost residual hearing immediately following surgery and was unable to use EAS. This subject was tested with the cochlear implant alone and is not included in this analysis.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of words correct (CUNY)
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 66
percentage of words correct (CUNY) | 42.2 (29.8)

2. Secondary Outcome: Improvement in Speech Perception in Noise With EAS When Compared to the Cochlear Implant Alone Condition
Description: CUNY sentences in noise are scored as the percent correct of words in each sentence. The total percent correct for the CI Alone condition was subtracted from the total percent correct for the EAS condition at 12 months giving an improvement in speech perception with EAS compared to CI Alone.
Time Frame: 12 months initial activation
Population: One subject lost residual hearing immediately after surgery and was unable to use EAS. The subject was testing in cochlear implant alone condition.
Measure: Mean (Standard Deviation); unit: percentage of words correct (CUNY)
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 66
percentage of words correct (CUNY) | 18.4 (22.03)

3. Secondary Outcome: Improvement on Speech Perception in the CI-only Condition as Compared to the Preoperative With Hearing Aid Condition.
Description: CNC words are scored as the percent correct out of 50 words. The percent correct for preoperative hearing aid use was subtracted from the percent correct for CI Alone at 12 months giving an improvement on speech perception for CI Alone compared to preoperative hearing aids.
Time Frame: 12 months post initial activation
Measure: Mean (Standard Deviation); unit: percentage of words correct (CNC)
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 67
percentage of words correct (CNC) | 18.0 (23.0)

4. Secondary Outcome: Increased Benefit With EAS as Compared to Their Preoperative Hearing Aid Condition as Measured by the APHAB Questionnaire.
Description: A lower score on the APHAB indicates a better performance. The global score for preoperative hearing aid use was subtracted from the global score for EAS at 12 months giving an improvement on the APHAB with EAS.
Time Frame: 12 months post initial activation
Population: Only 59 subjects completed the APHAB at preop and 12 months post activation.
Measure: Mean (Standard Deviation); unit: percentage of scoring change (APHAB)
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 59
percentage of scoring change (APHAB) | -30.2 (20.4)

5. Secondary Outcome: Increase in Satisfaction With EAS Compared to Preoperative Hearing Aid Condition as Measured by the HDSS.
Description: Satisfaction is ranked from 1-5, with 1 being very dissatisfied and 5 being very satisfied. Data reported is the percentage of subjects who experienced an increase in satisfaction when using EAS compared to preoperative hearing aids.
Time Frame: 12 months post initial activation
Population: Only 59 subjects completed the HDSS at preop and 12 month post activation.
Measure: Count of Participants; unit: Participants
Arm/Group | Original Audiological Criteria
Number analyzed (Participants) | 59
Participants | 51

ADVERSE EVENTS:
Arm/Group | Original Audiological Criteria
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 10/73
Other Adverse Events (participants affected / at risk) | 14/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Audiological Criteria (N=73)
Profound/total loss of residual hearing (Ear and labyrinth disorders) | 8 (8)
Electrode migration (Ear and labyrinth disorders) | 1 (1)
Electrode lead breakage (Ear and labyrinth disorders) | 1 (1) — Excess micro-movements caused by subject
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Audiological Criteria (N=73)
Type B/Type C tympanogram (Ear and labyrinth disorders) | 6 (8)
Conductive hearing loss (Ear and labyrinth disorders) | 5 (5)
Pain at implant site (Ear and labyrinth disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall not publish until after the multi center publication, provided that the multi center publication is submitted within 12 months after conclusion of the study.